CLINICAL TRIAL: NCT05286593
Title: Quantification of Myocardial Blood Flow by 3D Positron Emission Tomography With High and Low Rate Rb82 Infusion Profiles
Brief Title: 3D PET Myocardial Blood Flow and Rb82 Infusion Profiles
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ochsner Health System (Other)
Collaborators: Bracco Corporate (Industry)
Responsible Party: Principal Investigator, Robert Bober, M.D., Director of Nuclear Cardiology, Ochsner Health System
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00001584
Record Dates: First submitted 2021-12-29; First posted 2022-03-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Normal Healthy Volunteers Without Chronic Medical Conditions; Coronary Artery Disease; Cardiac Risk Factors; Myocardial Infarction
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: All participants will receive a standard "high flow rate" weight based bolus of Rb-82 and a "low flow rate" weight based infusion of Rb-82. The bolus and infusion doses will be administered randomly at rest and stress however the bolus is considered the gold standard.
  In addition, under resting conditions, participants will also receive a third dose of Rb-82 that is either a bolus or low flow rate (assigned randomly).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Normal volunteers (Other): Normal participants will receive serial doses of Rb-82 administered as either a bolus (B) (gold standard) or slow infusion (SI). Under resting conditions, they will receive 3 weight based doses. The first two doses are randomly assigned B and SI. The third dose is either B or SI. Under stress conditions, they will receive 2 weight based doses that are randomly assigned B and SI.
  Interventions: Drug: Slow Infusion of Rubidium-82
- Clinical patients (Other): Clinical patients participants will receive serial doses of Rb-82 administered as either a bolus (B) (gold standard) or slow infusion (SI). Under resting conditions, they will receive 3 weight based doses. The first two doses are randomly assigned B and SI. The third dose is either B or SI. Under stress conditions, they will receive 2 weight based doses that are randomly assigned B and SI.
  Interventions: Drug: Slow Infusion of Rubidium-82
- Infarcts (Other): Infarct participants will receive serial doses of Rb-82 administered as either a bolus (B) (gold standard) or slow infusion (SI). Under resting conditions, they will receive 3 weight based doses. The first two doses are randomly assigned B and SI. The third dose is either B or SI. Under stress conditions, they will receive 2 weight based doses that are randomly assigned B and SI.
  Interventions: Drug: Slow Infusion of Rubidium-82

INTERVENTIONS:
Drug: Slow Infusion of Rubidium-82 — Normal volunteers will receive weight based doses of Rb-82 infused as a slow infusion
  Other Names: 20 mls/min of Rubidium-82
  Arms: Normal volunteers
Drug: Slow Infusion of Rubidium-82 — Clinical patients will receive weight based doses of Rb-82 infused as a slow infusion
  Other Names: 20 mls/min of Rubidium-82
  Arms: Clinical patients
Drug: Slow Infusion of Rubidium-82 — Infarct volunteers will receive weight based doses of Rb-82 infused as a slow infusion
  Other Names: 20 mls/min of Rubidium-82
  Arms: Infarcts

SUMMARY:
The investigators seek to test bolus infusions (50ml/min) vs. slow infusions (20 ml/min) of Rb-82 on metrics of coronary blood flow assessed on a modern 3D PET/CT.

DETAILED DESCRIPTION:
As perfusion metrics in the healthy volunteers, patients with risk factors and/or coronary artery disease and in tissue with transmural myocardial infarctions has been well defined AND same day test-retest variability minutes apart using a bolus infusion is ±10%, the investigators shall test 3 hypotheses. The first hypothesis is repeated same day test-retest coefficient of variation (COV) of whole heart rMBF and sMBF acquired using a bolus infusion profile (50 mls/min) on a modern 3D PET scanner falls within ± 10%. The second hypothesis is repeated same day test-retest COV of whole heart rMBF and sMBF acquired using a slow infusion activity profile (20 mls/min) on a modern 3D PET scanner falls within ± 10%. The third hypothesis is COV of whole heart rMBF and sMBF between bolus and slow activity profiles is ± 10% where the bolus is considered the standard on a modern 3D PET scanner.

The investigators will test the different activity profiles on 3 distinct populations:

1. Healthy volunteers
2. Clinical volunteers with risk factors and/or CAD
3. Volunteers with clinical infarcts.

ELIGIBILITY:
Inclusion Criteria:

Normal Volunteers

* Adults ≥18 and <40 years old able to give informed consent.
* Ability to abstain from caffeine for 48 hours

The "clinical" population

* Adults ≥18 years old able to give informed consent.
* Any cardiac risk factor including hypertension, hyperlipidemia, diabetes mellitus or tobacco use OR
* CAD defined by with history of PCI or CABG, Coronary Ca score>400, or dense coronary calcifications noted on chest CT
* Ability to abstain from caffeine for 48 hours

The "infarct" population

* Adults ≥18 years old able to give informed consent.
* Prior cardiac PET scan demonstrating a fixed defect ≥ 15% of the LV myocardium with relative uptake ≤60% maximum uptake.
* In addition, to the perfusion defect, each volunteer requires either:

  * FDG PET or MRI viability studies confirming infarct OR
  * akinesis and wall thinning on ECHO within the same territory as the PET defect in addition to Q-waves on ECG
* Ability to abstain from caffeine for 48 hours

Exclusion Criteria:

Normal Volunteers

* Any chronic cardiac disease or condition (e.g., hypertension, hyperlipidemia)
* Any chronic systemic disease or condition (e.g., diabetes, systemic lupus, rheumatoid arthritis)
* Tobacco use
* Family history in a first degree relative with clinical CAD (h/o PCI, MI or CABG) in men <55 or women <65
* Severe claustrophobia
* Positive urine pregnancy test
* Inability to give informed consent
* BMI ≥ 30 or BMI>25 and <30 provided waist to hip ratio >0.80 in women or 0.90 in men.

The "clinical" and "infarct" populations

* Severe claustrophobia
* Hemodynamic instability or unstable symptoms
* Positive urine pregnancy test
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Resting and stress whole heart myocardial blood flow using the bolus infusion profile of Rubidium-82 | 1 day
  resting and stress myocardial blood flow in cc/min/g

SECONDARY OUTCOMES:
Resting and stress whole heart myocardial blood flow using the slow infusion profile of Rubidium-82 | 1 Day
  resting and stress myocardial blood flow in cc/min/g

CONTACTS AND LOCATIONS:
Locations (1):
- Ochsner, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Araujo LI, Lammertsma AA, Rhodes CG, McFalls EO, Iida H, Rechavia E, Galassi A, De Silva R, Jones T, Maseri A. Noninvasive quantification of regional myocardial blood flow in coronary artery disease with oxygen-15-labeled carbon dioxide inhalation and positron emission tomography. Circulation. 1991 Mar;83(3):875-85. doi: 10.1161/01.cir.83.3.875. PMID 1900224
- [Background] Bergmann SR, Fox KA, Rand AL, McElvany KD, Welch MJ, Markham J, Sobel BE. Quantification of regional myocardial blood flow in vivo with H215O. Circulation. 1984 Oct;70(4):724-33. doi: 10.1161/01.cir.70.4.724. PMID 6332687
- [Background] Sdringola S, Johnson NP, Kirkeeide RL, Cid E, Gould KL. Impact of unexpected factors on quantitative myocardial perfusion and coronary flow reserve in young, asymptomatic volunteers. JACC Cardiovasc Imaging. 2011 Apr;4(4):402-12. doi: 10.1016/j.jcmg.2011.02.008. PMID 21492816
- [Background] Renaud JM, DaSilva JN, Beanlands RS, DeKemp RA. Characterizing the normal range of myocardial blood flow with (8)(2)rubidium and (1)(3)N-ammonia PET imaging. J Nucl Cardiol. 2013 Aug;20(4):578-91. doi: 10.1007/s12350-013-9721-3. Epub 2013 May 9. PMID 23657833
- [Background] Merlet P, Mazoyer B, Hittinger L, Valette H, Saal JP, Bendriem B, Crozatier B, Castaigne A, Syrota A, Rande JL. Assessment of coronary reserve in man: comparison between positron emission tomography with oxygen-15-labeled water and intracoronary Doppler technique. J Nucl Med. 1993 Nov;34(11):1899-904. PMID 8229231
- [Background] Kern MJ, Bach RG, Mechem CJ, Caracciolo EA, Aguirre FV, Miller LW, Donohue TJ. Variations in normal coronary vasodilatory reserve stratified by artery, gender, heart transplantation and coronary artery disease. J Am Coll Cardiol. 1996 Nov 1;28(5):1154-60. doi: 10.1016/S0735-1097(96)00327-0. PMID 8890809
- [Background] Gewirtz H, Fischman AJ, Abraham S, Gilson M, Strauss HW, Alpert NM. Positron emission tomographic measurements of absolute regional myocardial blood flow permits identification of nonviable myocardium in patients with chronic myocardial infarction. J Am Coll Cardiol. 1994 Mar 15;23(4):851-9. doi: 10.1016/0735-1097(94)90629-7. PMID 8106689
- [Background] Rivas F, Cobb FR, Bache RJ, Greenfield JC Jr. Relationship between blood flow to ischemic regions and extent of myocardial infarction. Serial measurement of blood flow to ischemic regions in dogs. Circ Res. 1976 May;38(5):439-47. doi: 10.1161/01.res.38.5.439. PMID 1269083
- [Background] Kitkungvan D, Johnson NP, Roby AE, Patel MB, Kirkeeide R, Gould KL. Routine Clinical Quantitative Rest Stress Myocardial Perfusion for Managing Coronary Artery Disease: Clinical Relevance of Test-Retest Variability. JACC Cardiovasc Imaging. 2017 May;10(5):565-577. doi: 10.1016/j.jcmg.2016.09.019. Epub 2016 Dec 21. PMID 28017383
- [Background] Murthy VL, Bateman TM, Beanlands RS, Berman DS, Borges-Neto S, Chareonthaitawee P, Cerqueira MD, deKemp RA, DePuey EG, Dilsizian V, Dorbala S, Ficaro EP, Garcia EV, Gewirtz H, Heller GV, Lewin HC, Malhotra S, Mann A, Ruddy TD, Schindler TH, Schwartz RG, Slomka PJ, Soman P, Di Carli MF, Einstein A, Russell R, Corbett JR. Clinical Quantification of Myocardial Blood Flow Using PET: Joint Position Paper of the SNMMI Cardiovascular Council and the ASNC. J Nucl Cardiol. 2018 Feb;25(1):269-297. doi: 10.1007/s12350-017-1110-x. No abstract available. PMID 29243073
- [Background] Renaud JM, Yip K, Guimond J, Trottier M, Pibarot P, Turcotte E, Maguire C, Lalonde L, Gulenchyn K, Farncombe T, Wisenberg G, Moody J, Lee B, Port SC, Turkington TG, Beanlands RS, deKemp RA. Characterization of 3-Dimensional PET Systems for Accurate Quantification of Myocardial Blood Flow. J Nucl Med. 2017 Jan;58(1):103-109. doi: 10.2967/jnumed.116.174565. Epub 2016 Aug 18. PMID 27539843
- [Background] Bui L, Kitkungvan D, Roby AE, Nguyen TT, Gould KL. Pitfalls in quantitative myocardial PET perfusion II: Arterial input function. J Nucl Cardiol. 2020 Apr;27(2):397-409. doi: 10.1007/s12350-020-02074-8. Epub 2020 Mar 3. PMID 32128675
- [Background] Gould KL, Bui L, Kitkungvan D, Patel MB. Reliability and Reproducibility of Absolute Myocardial Blood Flow: Does It Depend on the PET/CT Technology, the Vasodilator, and/or the Software? Curr Cardiol Rep. 2021 Jan 22;23(3):12. doi: 10.1007/s11886-021-01449-8. PMID 33483794
- [Derived] Bober RM, Milani RV, Kachur SM, Morin DP. Assessment of resting myocardial blood flow in regions of known transmural scar to confirm accuracy and precision of 3D cardiac positron emission tomography. EJNMMI Res. 2023 Sep 27;13(1):87. doi: 10.1186/s13550-023-01037-7. PMID 37752344
- See also: Quantification of Resting Myocardial Blood Flow Using Rubidum82 Positron Emission Tomography in Regions with MRI-Confirmed Myocardial Scar. Annals of Nuclear Cardiology. — https://doi.org/10.17996/anc.21-00137

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/93/NCT05286593/Prot_SAP_000.pdf